CLINICAL TRIAL: NCT01175499
Title: Accuracy of Endoscopic Diagnosis of Carcinoma of the UpperAerodigestive Tract: A Tandem Trial of Direct Rigid Endoscopy and Transnasal Flexible Endoscopy With Narrowband Imaging
Brief Title: Concordance of Two Endoscopic Procedures for Diagnosis of Carcinoma of the Upper Aerodigestive Tract
Acronym: TNFE-NBI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to obtain funding to continue recruitment; no accrual
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 10-00166; 10201 (Other: UCSF Helen Diller Family Comprehensive Cancer Center)
Record Dates: First submitted 2010-07-20; First posted 2010-08-04 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Upper Aerodigestive Tract Lesions; Neoplasms, Oropharyngeal; Oropharyngeal Cancer; Neoplasms, Hypopharyngeal; Hypopharyngeal Cancer; Head and Neck Neoplasms; UADT Neoplasms; Carcinoma, Squamous Cell; Papilloma
Keywords: laryngoscopy; Laryngoscopic Surgery; laryngoscopes; upper aerodigestive tract lesions; endoscopy; biopsy
MeSH Terms: conditions — Oropharyngeal Neoplasms; Hypopharyngeal Neoplasms; Head and Neck Neoplasms; Carcinoma, Squamous Cell; Papilloma | interventions — Narrow Band Imaging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Direct Rigid Endoscopy — Laryngoscopy is performed under general anesthesia with a rigid laryngoscope. Mucosal surfaces of the oropharynx, hypopharynx, and glottis (base of tongue, vallecula, epiglottis, aryepiglottic folds, arytenoids, piriform sinuses, true and false vocal cords, and esophageal inlet) are systematically visualized. Areas of irregularity are biopsied with 2mm and/or 4mm cupped forceps. Esophagoscopy and bronchoscopy will be performed per the standard of care.
  Other Names: Rigid laryngoscope
Device: Transnasal Flexible Endoscopy with Narrowband Imaging — Transnasal flexible endoscopy with and without narrowband imaging- additional diagnostic test. This examination is performed after topical intranasal anesthesia with 2% Pontocaine spray. A fiberoptic laryngoscope is passed into the nasal cavity to the pharynx where mucosal surfaces of the UADT can be visualized. The optics of a standard fiberoptic scope are generally considered to be inferior to direct visualization. The addition of narrowband imaging does not change the procedure, but enhances visualization of the mucosal vasculature. Biopsies are performed through a second channel in the endoscope with 1.8mm cupped forceps and will require an additional dose of topical anesthesia.
  Other Names: EVIS EXERA 160A System

SUMMARY:
This study will compare TNFE-NBI and biopsy, with DRE and biopsy for the diagnostic evaluation and staging of patients with suspicious UADT lesions. All patients enrolled in the study will undergo TNFE-NBI with biopsy of suspicious lesions prior to planned regular clinical care (DRE). Biopsies will be evaluated by standard clinical methods for patient diagnoses and care. As the current standard of care, if all biopsies for a given patient are non-malignant, a 3 month office visit will be arranged to evaluate and determine the need for further intervention. At the end of study enrollment both sets of biopsies will be re-evaluated in a blinded fashion by the surgical pathologist. Study assessment of malignant vs. non-malignant (benign) pathology will be used to see whether both tests tended to agree on diagnoses.

DETAILED DESCRIPTION:
This is a single arm prospective study to evaluate the concordance between a standard-of-care diagnostic procedure and TNFE-NBI for diagnosing malignancy. The primary aim of this investigation is to determine whether the TNFE NBI procedure can detect and stage cancer in the head and neck as well as the standard DRE which requires general anesthesia.

Patients who are pending direct laryngoscopy after presenting to the Department of Otolaryngology-Head and Neck Surgery at UCSF with UADT lesions will be asked to participate in the study provided all eligibility criteria are met. Under current standard-of-care for diagnostic evaluation and staging of UADT lesions, patients will undergo imaging studies including CT and/or MRI of the neck with contrast prior to direct laryngoscopy. Study participants will undergo both the TNFE NBI and DRE procedures.

The study procedure TNFE NBI will be performed, followed 1-6 weeks later by DRE, the standard approach for diagnosis, without the surgeon having knowledge of the details of the first procedure. The sequence of examinations in this investigation is dictated by the need to minimize mucosal trauma during the first examination and allow for mucosal healing prior to the second examination, and thus cannot be randomized. TNFE-NBI produces much less mucosal trauma by avoiding direct blunt manipulation and through the smaller, 1.8mm, cupped biopsy forceps.

Because it is possible that the TNFE NBI procedure might detect smaller tumors or lesions in different locations, the biopsy locations from the TNFE NBI procedure will be made known at the end of the DRE surgery to ensure that all needed areas are biopsied. Therefore, a secondary aim of this study will be to explore whether the TNFE NBI procedure may improve the detection of malignancy when added to the DRE surgery.

Patients enrolling in the study will undergo TNFE-NBI with biopsy of suspicious lesions. The TNFE-NBI examinations will be digitally recorded. The examiner will describe, using standard language and diagrams, anatomic location of suspicious areas revealed during the procedure. Biopsy tissue will be labeled as to the area of origin.

In the event that a participant does not tolerate TNFE-NBI, the study procedure will be aborted.

At least one week and no more than 6 weeks after TNFE-NBI, patients will undergo standard of care direct rigid endoscopy. The intervening time to DRE is to allow for recovery of mucosal surfaces.

Participants who did not tolerate TNFE-NBI will undergo DRE as standard of care.

The DRE examiner will be blinded as to which areas were biopsied during the TNFE-NBI procedure until completion of the standard of care DRE examination and tissue biopsy selection. In the investigator's experience, areas of prior biopsy will not be apparent to the DRE examiner as mucosal recovery will occur during 1-6 weeks elapsing between TNFE-NBI and DRE. Upon completion of the standard of care DRE examination and tissue biopsy selection, the DRE examiner will open the TNFE-NBI examiner's note describing the areas deemed suspicious during TNFE-NBI. Additional areas may then be examined and biopsied with DRE based on the TNFE-NBI note. Records will be kept as to which anatomic areas were:

1. identified by both procedures,
2. identified by DRE only after prompting by the TNFE-NBI note
3. identified by DRE only (not previously identified by TNFE-NBI).

A diagnosis of carcinoma in situ or invasive squamous cell carcinoma will be considered positive for malignancy. If a diagnosis of malignancy is made after the initial endoscopy, regardless of which test was positive, the patient will be contacted immediately so that appropriate treatment can be pursued. For diagnoses of dysplasia and other non-malignant conditions such as polyp, lymphoid tissue, papilloma, etc., the patient will be scheduled for follow-up.

Routine follow-up of benign lesions includes a routine head and neck examination, including indirect laryngoscopy with a fiberoptic endoscope 2-3 months after biopsy. New or enlarging lesions will be assessed in the operating room with DRE per standard of care. Lesions initially diagnosed as non-malignant that are stable or not visualized at follow-up will not need re-biopsy per standard of care.

At the conclusion of study enrollment, all biopsy specimens will be de-identified, batched, and evaluated by a pathologist blinded to the type of endoscopy. A diagnosis of carcinoma in situ or invasive squamous cell carcinoma will be considered positive for malignancy.

If patients with non-malignant diagnoses of study pathology (both TNFE-NBI and DRE) have been diagnosed with malignancy at or before routine follow-up, the study evaluation will be considered a false negative. If no malignancy developed within three months of the biopsy procedures, the study evaluation will be considered a true negative. (This design represents a compromise in evaluating patients with a negative endoscopy. By necessity a negative diagnosis is one of exclusion, given that complete pathologic evaluation of every patients' upper aerodigestive tract is neither ethical, practical, nor feasible in clinical practice. Precedent for this design can be found in Smith-Bindman, Chu et al. 2005)

ELIGIBILITY:
Inclusion Criteria:

* Age eighteen years or older
* Patients who are pending operative direct laryngoscopy as standard clinical care
* Presence of upper aerodigestive tract (UADT) (oropharyngeal, hypopharyngeal and/or glottic mucosal) lesion(s) suspicious for diagnoses including but not limited to: squamous cell carcinoma, carcinoma in situ, squamous dysplasia, papilloma, OR presence of diagnosed metastatic squamous cell carcinoma in the neck with an unidentified primary lesion
* Ability to give written informed consent and willingness to comply with the requirements of the protocol

Exclusion Criteria:

* Patients who are not medically able to undergo TNFE
* Allergy to topical anesthesia
* Active lymphoma
* Lesion inaccessibility to TNFE: oral cavity (anterior 2/3 tongue, buccal mucosa)
* Coagulopathy: INR ≥ 1.5
* Any condition that compromises compliance with the objectives and procedures of this protocol, as judged by the principal investigator such as anxiety or narrow nasal passage way.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07

PRIMARY OUTCOMES:
Agreement between TNFE-NBI and DRE | Within approximately 6 weeks of enrollment, after both diagnostic procedures have been completed
  At the conclusion of study enrollment, all biopsy specimens will be coded, de-identified, and re-evaluated by the study pathologist in a blinded fashion. The code will be broken for the purposes of study analyses.
  If all biopsies taken by both procedures on each patient are diagnosed as non-malignant upon blinded evaluation by the study pathologist or if both procedures have at least one biopsy diagnosed as malignant, this will be considered concordance.

SECONDARY OUTCOMES:
Agreement of TNFE-NBI and DRE on tumor stage and location | Within approximately 6 weeks of enrollment, after both diagnostic procedures have been completed
  Describe differences, if any, in characterization of AJCC cTNM stage and tumor location as determined by TNFE-NBI as compared to standard-of-care DRE
Agreement between TNFE-NBI and DRE on biopsy location selection | Within approximately 6 weeks of enrollment, after both diagnostic procedures have been completed
  describe differences, if any, in biopsy location during TNFE-NBI as compared to standard-of-care DRE
False negative diagnoses by TNFE-NBI or DRE | Approximately 4 months after enrollment, after completion of both procedures and 3-month follow-up for non-malignant diagnoses
  To describe the frequency of detecting malignancy at a 3-month follow-up for patients initially diagnosed as negative for malignancy by both TNFE NBI and DRE evaluations
Frequency and Timing of Adverse Events | Within approximately 6 weeks of enrollment, after both diagnostic procedures have been completed and patient follow-up at 30 days
  The frequency by grade for all adverse events will be tabulated by type and procedure as well as timing (during or immediately following study procedure vs. follow-up).
Describe patient tolerance for TNFE-NBI | At the time of TNFE-NBI procedure, study day 1
  Patients who have fulfilled the inclusion criteria and are unable to tolerate the unsedated examination will be classified as having non-concordance between TNFE-NBI and DRE (because a diagnosis could not be made based upon pathology) and the reason for intolerance to the procedure recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Mark S. Courey, MD, Principal Investigator — UCSF Helen Diller Family Comprehensive Cancer Center, Otolaryngology, Head & Neck Surgery